CLINICAL TRIAL: NCT04362709
Title: A Prospective Cohort Study of Post-anesthesia Management in Patients Undergoing Neurosurgery
Brief Title: Study of Post-anesthesia Management in Patients Undergoing Neurosurgery
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Associate professor, Beijing Tiantan Hospital
Other Study IDs: 2019-10
Record Dates: First submitted 2020-01-14; First posted 2020-04-27 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Neurosurgery; Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative complications
- No postoperative complications

SUMMARY:
The postoperative complications of neurosurgery are various and complex, which brings heavy economic and social burden to families. Timely detection and early intervention can help reduce the incidence of adverse events and mortality. The main purpose of this study is to analyze the possible factors related to postoperative complications of Neurosurgery, so as to achieve the prospective prevention and treatment of postoperative complications of neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients received neurosurgery in Beijing Tiantan hospital.

Exclusion Criteria:

* Preoperative severe cognitive dysfunction ；
* Refused to sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients expected to returned to post-anesthesia care unit(PACU) after neurosurgical treatment in Beijing Tiantan hospital.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2028-11-22 (Estimated); Study Completion 2028-11-22 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative complications in neurosurgery. | 5±2 days
  The incidence of postoperative complications was diagnosed by the corresponding assessment scale.Complications include nausea, vomiting, delirium, delayed recovery, intracranial hematoma,etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, M.D., Ph.D, Study Chair — Department of Anesthesiology, Beijing Tiantan Hospital
Locations (1):
- Beijing TianTan Hospital, Beijing, China